CLINICAL TRIAL: NCT00055718
Title: A Pilot Study of Silymarin During Maintenance Therapy in Children With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Silymarin (Milk Thistle Extract) in Treating Patients With Acute Lymphoblastic Leukemia Who Are Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000270914; CPMC-IRB-14117
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2006-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Leukemia
Keywords: drug/agent toxicity by tissue/organ; childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Silymarin

INTERVENTIONS:
Dietary Supplement: silymarin

SUMMARY:
RATIONALE: Silymarin (milk thistle extract) is an herb that may be effective in treating liver disorders caused by cancer therapy.

PURPOSE: Randomized phase II trial to study the effectiveness of silymarin in treating patients who have acute lymphoblastic leukemia with chemotherapy-related side effects to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of silymarin, in terms of liver function tests, in patients with acute lymphoblastic leukemia receiving hepatotoxic chemotherapy.
* Determine the effect of this drug on free and conjugated serum silibinin values in these patients.
* Determine the serum antioxidant capacity by Oxygen Radical Absorbance Capacity in patients treated with this drug.
* Determine the oxidative damage, as determined by 8-oxodeoxyguanosine adducts, in patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral silymarin daily for 28 days.
* Arm II: Patients receive oral placebo as in arm I. Patients are followed at day 56.

PROJECTED ACCRUAL: A total of 50 patients (25 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)
* Currently receiving maintenance or continuation phase chemotherapy for ALL

  * Regimen comprising intrathecal and oral methotrexate; vincristine IV; oral prednisone or dexamethasone; and oral mercaptopurine
* Elevated liver function tests, evidenced by 1 of the following criteria:

  * Bilirubin greater than 1.5 times upper limit of normal (ULN)
  * AST greater than 2.5 times ULN
  * ALT greater than 2.5 times ULN

PATIENT CHARACTERISTICS:

Age

* 2 to 21

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* See Disease Characteristics

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-11; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Effect of silymarin on elevated liver function tests (AST, ALT, total bilirubin, and direct bilirubin) at baseline, day 28, and day 56

SECONDARY OUTCOMES:
Serum antioxidant capacity as measured by the Oxygen Radical Absorbance Capacity (ORAC) at baseline, day 28, and day 56
Oxidative damage as measured by 8-oxodeoxyguanosine adducts at baseline, day 28, and day 56

CONTACTS AND LOCATIONS:
Overall Officials: Kara Kelly, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (8):
- United States (7):
  - Miami Children's Hospital, Miami, Florida
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Ladas EJ, Kroll DJ, Oberlies NH, Cheng B, Ndao DH, Rheingold SR, Kelly KM. A randomized, controlled, double-blind, pilot study of milk thistle for the treatment of hepatotoxicity in childhood acute lymphoblastic leukemia (ALL). Cancer. 2010 Jan 15;116(2):506-13. doi: 10.1002/cncr.24723. PMID 20014183